CLINICAL TRIAL: NCT02324439
Title: Flaxseed as Maintenance Therapy for Ovarian Cancer Patients in Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Brard-SIUSOM-2014-004
Record Dates: First submitted 2014-11-21; First posted 2014-12-24 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: ovarian cancer; flaxseed; dietary supplement; organic dietary supplement; recurrence
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega Nutrition cold-milled flaxseeds (Experimental): All subjects will receive a 20g daily dose of cold-milled flaxseeds for 24 months.
  Interventions: Drug: Omega Nutrition cold-milled flaxseeds

INTERVENTIONS:
Drug: Omega Nutrition cold-milled flaxseeds — Patients who are currently in clinical remission will receive a daily 20g dose of cold milled flaxseed as a dietary supplement to determine if this intervention prolongs clinical remission.
  Other Names: cold-milled flaxseeds

SUMMARY:
This is a phase 0/phase I feasibility trial to test the hypothesis that flaxseed supplementation is an effective maintenance therapy for patients with ovarian cancer who are in clinical remission following platinum-based regimens. The investigators further hypothesize levels of estrogen metabolites and prostaglandin E2 in this patient population will correlate with recurrence of disease, extent of tumor burden, invasion and metastasis.

DETAILED DESCRIPTION:
For the year 2014, it is projected there will be 21,980 women diagnosed and 14,270 deaths from ovarian cancer (OC) in the US. OC is the leading cause of death from gynecologic malignancies and ranks second among newly diagnosed gynecological cancers in the United States. More than 70% of patients present with advanced disease (stages II-IV). Although most patients (70-80%) initially respond to cytoreductive surgery and adjuvant paclitaxel and platinum-based chemotherapy, approximately 80% of these women will experience disease recurrence. For stages III and IV, the risk of recurrence is very high, with 5-year survival rates ranging from just 13% to 44%. Furthermore, OC represents a high potential for metastases even in the setting of complete response to initial therapy. Efforts to devise new treatment strategies are therefore essential in order to improve survival. In this grant application, the investigators postulate that utilizing dietary supplementation of flaxseed for maintenance therapy in patients with OC in clinical remission following treatment with platinum-based regimens will be tolerable and prolong their progression-free survival (PFS). The investigators hypothesis is based on the following:

* Data from the investigators laboratory revealed that flaxseed effectively decreased severity and progression of OC in the only spontaneous preclinical egg-laying hen model that fully recapitulates human OC.
* In a phase II study, flaxseed supplementation reduced proliferation rates of prostate cancer after just 30 days.
* Flaxseed has been shown to inhibit solid tumor growth and metastases in several other preclinical cancer models (breast, prostate, colon).
* Flaxseed is a safe dietary supplement for cancer patients.
* Flaxseed supplementation increased survival in our investigators' animal model and these flaxseed-fed hens exhibited lower inflammatory markers and maintained a healthy weight, inferring a better quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of OC including epithelial ovarian carcinoma, primary peritoneal cancer or fallopian tube cancer who are currently in clinical remission as determined by the PI or co-I and are within 4 months of completion of cancer treatment.
* Patients at risk of clinical relapse: patients of any stage who are in remission who have undergone surgical debulking and adjuvant chemotherapy.
* Patients must have adequate:

  * Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to Common Toxicity Criteria (CTCAE v4.0) Grade 1. Platelets greater than or equal to 100,000/mcl (CTCAE v4.0 Grade 0-1). Hemoglobin (Hgb) greater than or equal to 9.0g/dl (CTCAE v4.0 Grade 2).
  * Renal function: Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v4.0 Grade 1.
  * Hepatic function: Bilirubin less than or equal to 1.5 x ULN (CTCAE v4.0 Grade 1). Serum glutamate oxaloacetate transaminase (SGOT) and alkaline phosphatase ≤ 2.5 x ULN (CTCAE v4.0 Grade 1).
* Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients with ovarian cancer of low malignant potential (borderline cancers).
* Patients who have received prior radiotherapy or chemotherapy for another malignancy.
* Patients who are pregnant or lactating.
* Patients with serious medical or psychiatric illness.
* Patients with a history of inflammatory bowel disease, problems with chronic diarrhea or history of bowel obstruction.
* Patient has received other investigational drugs within 28 days before enrollment.
* Patients with concurrent uncontrolled illness.
* Patients unable to tolerate and/or allergies to flaxseed or flaxseed preparations.
* Patients with Gynecologic Oncology Group (GOG) performance status > 2.
* Patients with a history of uncontrolled diabetes (as flaxseed can lower blood glucose levels and might have additive effects when used with anti-diabetic drugs).
* Patients concurrently using anticoagulants/antiplatelets on a DAILY BASIS, including aspirin, Clopidogrel (Plavix), Ticlopidine (Ticlid), and Coumadin.
* Patients with a diagnosis of/problems with von Willebrand's disease or other bleeding disorders (as flaxseed may slow blood clotting; the risk of bruising or bleeding in people on anticoagulants or with bleeding disorders may be a concern).
* Flaxseed supplementation may be contraindicated in patients with acute abdomen, esophageal stricture or perforation, dysphagia, GI obstruction or ileus, acute intestinal inflammation or unexplained abdominal pain. Patients with any of these conditions will be excluded from this trial as the high fiber content of flaxseed may make these conditions worse

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of consuming 20g of flaxseed per day | 24 months
  To determine the feasibility of administering a 20 gram (g) per day dose of ground flaxseed to patients with histology-proven epithelial ovarian cancer who have undergone surgical debulking and adjuvant chemotherapy with platinum-based regimens and are currently in clinical remission.

SECONDARY OUTCOMES:
Progression free survival (PFS) | change from baseline values over 24 months
  Analysis of CA-125, review of symptoms and imaging (if indicated)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brard, MD, PhD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States